CLINICAL TRIAL: NCT06502886
Title: Evaluation of The Stability of Orthodontic Treatment After First Premolar Extraction in Adult Patients Using Bonded Retainer Versus Bonded Retainer Combined With Vacuum Formed Retainer : A Randomized Clinical Trial
Brief Title: Evaluation of The Stability of Orthodontic Treatment After First Premolar Extraction Using Combined Retention Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelaziz Taha Abdelaziz Malek, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ORTH 3-3-10
Record Dates: First submitted 2024-06-30; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blinded randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): Use bonded retainer combined with vacuum formed retainer
  Interventions: Procedure: combined protocol of retention (bonded lingual retainer and vacuum formed retainers)
- The comparator group (Active Comparator): Use bonded retainer
  Interventions: Procedure: Bonded lingual retainer

INTERVENTIONS:
Procedure: combined protocol of retention (bonded lingual retainer and vacuum formed retainers) — Combined bonded retainer and vacuum formed retainer
  Other Names: Fixed lingual retainer and vacuum formed retainer
  Arms: The intervention group
Procedure: Bonded lingual retainer — Bonded retainer
  Other Names: Fixed lingual retainer
  Arms: The comparator group

SUMMARY:
The aim of this study is to compare between the stability of anterior and posterior segments in both arches using bonded lingual retainers versus a combined protocol of retention (bonded lingual retainer and vacuum formed retainers). The effect of different treatment changes achieved on the post-treatment stability will be studied in both groups.

Hypothesis: No difference between BR and BR+VFR regarding the stability of anterior segment alignment and posterior segment alignment and interdigitation

DETAILED DESCRIPTION:
Retention is necessary to be done after orthodontic treatment. It aids to prevent the tendency for relapse of teeth toward their pretreatment position. Fixed or removable retention appliances can reduce the risk of relapse, but to date there is still limited evidence on treatment protocols, wearing time and duration. However, long-term retention with bonded lingual retainers is commonly recommended and often considered the gold standard (method of first choice) in orthodontic retention. Regardless of the expected benefits concerning tooth stabilization, aesthetic appearance and independency from the patient's compliance, there have been increasing numbers of reports on undesirable changes in tooth position in the presence of retainers. Since "active" lingual retainers are able to exert forces to teeth, they have been suspected of causing torque changes of adjacent incisors ("X-effect"). Therefore, several authors recommend to insert removable and fixed in both arches for maximum relapse prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients at the end of comprehensive orthodontic treatment after extraction of upper and lower first premolars and requiring subsequent application of a lingual and palatal bonded retainers
2. Good oral hygiene
3. Patients whom the pre-treatment records (models) are available
4. Good finishing criteria (ABO grading system)

Exclusion Criteria:

1. Non-extraction orthodontic treatment
2. Poor oral hygiene
3. Dental/congenital anomalies ex: Missing laterals, transposed canines, Cleft lip and palate/craniofacial syndromes
4. Poor finishing criteria (ABO grading system)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Mandibular anterior segment alignment | 6 months
  Using 3D models, mandibular anterior segment alignment will be measured by little irregularity index

SECONDARY OUTCOMES:
Maxillary anterior segment alignment | 6 months
  Using 3D models, maxillary anterior segment alignment will be measured by little irregularity index

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medicine, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
All the members of the research team will have access to the study data. All the data will be secured to maintain confidentiality. No other parties are allowed to assess the results until the study is terminated and the conclusions are revealed.